CLINICAL TRIAL: NCT04893265
Title: Getting Asian Americans INFORMED to Facilitate COVID-19 Testing and Vaccination
Acronym: INFORMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Chinese Community Health Resource Center (Other); University of California, Davis (Other); University of California, Merced (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-32933; 3R01DA036749-05S1 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-19 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Educational Activities
Keywords: COVID-19 Testing; COVID-19 Vaccination; Asian Americans; Peer Education; Immigrants; Chinese American; Hmong American; Vietnamese American

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Messaging Only (Active Comparator): Participants will receive a weekly SMS Text or instant message on a topic related to COVID-19 testing over 12 weeks. In addition, participants will receive as-needed messages on updates of COVID-19 testing related information. The messages will be responsive to the rapid evolving developments and changes related to COVID-19 testing guidelines. Some of the messages will include a link to allow participants to get to the entire message/information on the study website.
  Interventions: Behavioral: Text Messaging Only
- INFORMED (Experimental): Participants will receive a weekly SMS Text or instant message on a topic related to COVID-19 testing as described in the "Text Messaging Only." In addition, participants will receive a Lay Health Worker (LHW) Educational Outreach Program, which includes 2 group sessions via video calls like Zoom or another video conferencing platform and 2 follow-up contacts via telephone, text or other media assignment.
  Interventions: Behavioral: INFORMED

INTERVENTIONS:
Behavioral: Text Messaging Only — Active Comparator
  Arms: Text Messaging Only
Behavioral: INFORMED — Experimental
  Arms: INFORMED

SUMMARY:
This study develops and evaluates the "INdividual and Family-Oriented Responsive Messaging EDucation" (INFORMED) intervention in increasing knowledge about COVID-19 testing and decreasing decisional conflicts of getting tested for COVID-19. A 2-arm randomized controlled trial will compare INFORMED delivered by LHW educational outreach plus Short Message Service (SMS) text messaging to SMS text with LHW support.

DETAILED DESCRIPTION:
This project "Getting Asian Americans INFORMED to Facilitate COVID-19 Testing and Vaccinations" is to identify and address sociocultural, ethical and behavioral barriers related to Coronavirus Disease 2019 (COVID-19) testing and vaccination to enable Asian Americans to make well-informed decisions about getting tested for COVID-19. Asian Americans have experienced high rates of COVID-19 related hospitalization and mortality rates when compared to non-Hispanic whites particularly among those who tested positive. Excess COVID-19 related deaths observed in Asian Americans are in part due to under-testing or delayed testing. Asian Americans may face multiple challenges, including sociocultural (limited English proficiency, lack of trust, excess fears and social stigma related COVID-19), ethical (lack of proven benefits of various guidelines, unequal access to testing resources), and behavioral (tobacco and e-cigarette use, other competitive behaviors) factors. The pandemic is rapidly evolving and presents urgent needs to develop highly efficient channels to communicate accurate, easily comprehensive, cultural appropriate and practical information. This application is a supplement to a parent R01 "A Family-Focused Intervention for Asian American Male Smokers," as known to the public as a community-based intervention research program "Healthy Family Project." Leveraging the community partnerships and the individual / family-based LHW intervention approaches developed by the study team, the proposed aims are: (1)Develop and evaluate "INdividual and Family-Oriented Responsive Messaging EDucation" (INFORMED) intervention in increasing knowledge about COVID-19 testing and decreasing decisional conflicts of getting tested for COVID-19. A 2-arm randomized controlled trial will compare INFORMED delivered by LHW educational outreach plus SMS text messaging to SMS text with LHW support. (2) Conduct in-depth prospective investigation of sociocultural, ethical and behavioral factors related to COVID-19 testing in Chinese, Hmong and Vietnamese American over-time. In addition, factors affecting acceptance for vaccination research trial participation and vaccination uptake and how vaccination acceptance is associated with COVID-19 testing uptake will be explored.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* self-identify as Chinese, Hmong or Vietnamese
* able to read and/or speak: English, Chinese (Cantonese/Mandarin), Hmong or Vietnamese;
* have access to a mobile phone to receive SMS text messages

Exclusion Criteria:

* unwilling to receive SMS text messages from the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Y Tsoh, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - The Fresno Center, Fresno, California
  - Chinese Community Health Resource Center, San Francisco, California
  - Immigrant Resettlement & Cultural Center Inc, San Jose, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and data use agreement must be signed.
Supporting Information: ICF
Time Frame: Approximately 9 months after data completion
Access Criteria: De-identified data will be shared upon request with a data use agreement.

REFERENCES:
- [Background] Cheng J, Tsoh JY, Guan A, Luu M, Nguyen IV, Tan R, Thao C, Yu E, Lor D, Pham M, Choi J, Kim M, Stewart SL, Burke NJ. Engaging Asian American Communities During the COVID-19 Era Tainted With Anti-Asian Hate and Distrust. Am J Public Health. 2022 Nov;112(S9):S864-S868. doi: 10.2105/AJPH.2022.306952. Epub 2022 Sep 15. No abstract available. PMID 36108257

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by 3 community-based agencies primarily through trained lay health workers.
Pre-assignment Details: Participants much complete baseline survey prior to randomization and assignment intervention groups. Participants could choose to participate as a dyad with another participant or participate individually. If the participants choose to participate as a dyad, both participants were randomized together in the same group. All data tables represent individual participants.
Period: Overall Study
Arm/Group | Text Messaging Only | INFORMED
Started | 121 | 126
Completed | 119 | 117
Not Completed | 2 | 9
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text Messaging Only | INFORMED | Total
Number analyzed (Participants) | 121 | 126 | 247
Age, Categorical [Count of Participants; unit: Participants] — Population: 6 participants with unknown age
  Participants
    number analyzed (Participants) | 119 | 122 | 241
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 98 | 111 | 209
    >=65 years | 21 | 11 | 32
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant did not provide sex
  Participants
    number analyzed (Participants) | 120 | 126 | 246
    Female | 71 | 77 | 148
    Male | 49 | 49 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 121 | 126 | 247
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 121 | 126 | 247
Participation mode [Count of Participants; unit: Participants] — Participants could choose to participate as a dyad with another participant, or to participate individually. If the participants choose to participate as a dyad both participants were randomized to the same treatment condition.
  Participants
    Individual | 63 | 68 | 131
    Dyad | 58 | 58 | 116
Education [Count of Participants; unit: Participants] — Categorical Population: 1 participant did not respond
  Participants
    number analyzed (Participants) | 120 | 126 | 246
    High School or Less/ Preferred Not to Answer | 55 | 45 | 100
    Some college/ Technical or Vocational School | 35 | 43 | 78
    Bachelor's Degree or Higher | 30 | 38 | 68
Marital Status [Count of Participants; unit: Participants] — Population: 7 participants did not respond
  Participants
    number analyzed (Participants) | 119 | 121 | 240
    Married/Living with Partner | 69 | 83 | 152
    Single/Preferred Not to Answer | 50 | 38 | 88
Household Description [Count of Participants; unit: Participants] — Population: 1 participant did not answer
  Participants
    number analyzed (Participants) | 120 | 126 | 246
    Family including kids | 67 | 66 | 133
    Multigenerational | 12 | 26 | 38
    No kids/Other | 41 | 34 | 75
Asian cultural groups [Count of Participants; unit: Participants]
  Chinese | 41 | 42 | 83
  Hmong | 40 | 44 | 84
  Vietnamese | 40 | 40 | 80
Nativity [Count of Participants; unit: Participants] — Population: 10 participants did not respond
  Participants
    number analyzed (Participants) | 118 | 119 | 237
    Born outside of United States | 86 | 93 | 179
    Born in the United States | 32 | 26 | 58
Years lived in the United States [Count of Participants; unit: Participants] — Population: 16 participants did not provide years lived in the U.S.
  Participants
    number analyzed (Participants) | 117 | 114 | 231
    10 or fewer | 26 | 26 | 52
    More than 10 (including U.S. born) | 91 | 88 | 179
Preferred Language [Count of Participants; unit: Participants]
  English | 69 | 74 | 143
  Non-English | 52 | 52 | 104
Self-rated Spoken English Proficiency [Count of Participants; unit: Participants] — Population: 1 participant did not respond
  Participants
    number analyzed (Participants) | 120 | 126 | 246
    Poorly/Not at all | 37 | 33 | 70
    So-so | 26 | 22 | 48
    Well/Fluently | 57 | 71 | 128
Health insurance [Count of Participants; unit: Participants] — Population: 3 participants did not respond
  Participants
    number analyzed (Participants) | 119 | 125 | 244
    Private Insurance | 45 | 64 | 109
    Other | 74 | 61 | 135
Employment status [Count of Participants; unit: Participants] — Population: 12 participants did not respond
  Participants
    number analyzed (Participants) | 119 | 116 | 235
    Currently working | 67 | 74 | 141
    Not currently working | 52 | 42 | 94
Self-rated Health [Count of Participants; unit: Participants] — Population: 4 participants did not respond
  Participants
    number analyzed (Participants) | 120 | 123 | 243
    Excellent/Very Good/Good | 99 | 109 | 208
    Fair/Poor/DK/NA | 21 | 14 | 35
Smoked cigarettes in the past 30 days [Count of Participants; unit: Participants] — Population: 4 participants did not respond
  Participants
    number analyzed (Participants) | 120 | 123 | 243
    No | 103 | 109 | 212
    Yes/DK/Preferred Not To Answer | 17 | 14 | 31
Getting Tested for COVID-19 in the Past Month [Count of Participants; unit: Participants] — Population: 3 participants did not respond
  Participants
    number analyzed (Participants) | 120 | 124 | 244
    No/Don't Know | 95 | 95 | 190
    Yes | 25 | 29 | 54
Intention to get tested for COVID-19 as often as needed [Count of Participants; unit: Participants] — Population: 3 participants did not respond
  Participants
    number analyzed (Participants) | 118 | 126 | 244
    No (do not agree) | 41 | 42 | 83
    Yes (agreed or strong agreed) | 77 | 84 | 161
Decisional Conflict of Getting Tested for COVID-19 ("SURE" test) [Mean (Standard Deviation); unit: units on a scale] — Decision conflict is measured by the 4-item Decision Making Conflict (SURE) test which asks whether participants: 1) know enough about benefits and harm; 2) clear about which benefits and harms matter most; 3) have enough support/advice to make a choice; and 4) feel sure about the best choice regarding getting tested for COVID-19. Each item is scored either 0 (unsure) or 1(sure). The total score ranges from 0 to 4. Higher scores indicate 'more sure,' lower scores indicate higher decisional conflict. Population: 5 participants did not respond
  units on a scale
    number analyzed (Participants) | 119 | 123 | 242
    (all) | 3.61 (0.86) | 3.55 (1.03) | 3.58 (0.95)
Getting a COVID-19 test is easy [Count of Participants; unit: Participants] — Population: 3 participants did not respond
  Participants
    number analyzed (Participants) | 119 | 125 | 244
    No (Do not agree) | 22 | 18 | 40
    Yes (Agree / strongly agree) | 97 | 107 | 204
Knew where to get COVID-19 testing [Count of Participants; unit: Participants] — Population: 4 participants did not respond
  Participants
    number analyzed (Participants) | 117 | 126 | 243
    No (Do not agree) | 28 | 21 | 49
    Yes (Agree / Strongly Agree) | 89 | 105 | 194
Knew of people in family or social network who had been tested for COVID-19 [Count of Participants; unit: Participants] — Population: 1 participant did not respond
  Participants
    number analyzed (Participants) | 120 | 126 | 246
    No | 15 | 13 | 28
    Yes | 105 | 113 | 218
Knowledge of COVID-19 test [Mean (Standard Deviation); unit: units on a scale] — The COVID-19 Test Knowledge Scale consists of 6 true-false items testing knowledge about interpretations related to positive or negative COVID-19 test results. The score is the sum of items that a participant answers correctly, ranged from 0 (no item was responded correctly) to 6 (all items were responded correctly).
  units on a scale | 4.58 (1.15) | 4.75 (0.98) | 4.67 (1.07)
Values about COVID-19 Testing [Mean (Standard Deviation); unit: units on a scale] — This is a 4-item scale asking participants to indicate their values or attitudes toward getting COVID-19 tested using on a 5-point scale (1 to 5) for each set of attributes: bad to good; unimportant to important; not reassuring to reassuring; a difficult decision to an easy decision. The scale score is computed by summing the score of all 4 items, ranged from 4 to 20. Population: 13 participants did not respond or complete the measure
  units on a scale
    number analyzed (Participants) | 116 | 118 | 234
    (all) | 18.33 (2.76) | 18.64 (2.02) | 18.48 (2.42)
COVID-19 cases per 1000,000 population [Mean (Standard Deviation); unit: cases per 100,000 population] — Number of COVID-19 cases per 100,000 population recorded within the past 30 days matched to individual participants' county of residence and time of baseline survey completion. Source of data: California Department of Public Health: COVID-19 Time-Series Metrics by County and State (ARCHIVED). Available at: https://data.chhs.ca.gov/dataset/covid-19-time-series-metrics-by-county-and-state.
  cases per 100,000 population | 846.08 (1261.78) | 890.75 (1441.03) | 868.87 (1353.62)

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict for Getting Tested for COVID-19
Description: Decision conflict is measured by the 4-item Decision Making Conflict (SURE) test which asks whether participants: 1) know enough about benefits and harm; 2) clear about which benefits and harms matter most; 3) have enough support/advice to make a choice; and 4) feel sure about the best choice regarding getting tested for COVID-19. Each item is scored either 0 (unsure) or 1(sure). The total score ranges from 0 to 4. Higher scores indicate 'more sure,' lower scores indicate higher decisional conflict.
Time Frame: Week 16
Population: Participants who completed the survey at Week 16 and provided all the information required to compute the variable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Only | INFORMED
Number analyzed (Participants) | 116 | 116
score on a scale | 3.89 (0.37) | 3.96 (0.24)
Statistical Analysis 1: Comparison: Text Messaging Only vs INFORMED; Test type: Superiority; p = 0.4471, Mixed Models Analysis; Mean Difference (Net) = 0.08540, 95% CI 2-sided [-0.1352 to 0.3060], Standard Error of Mean 0.1122

2. Secondary Outcome: Tested for COVID-19 During the Past Month
Description: Participants are asked to self-report whether they have been tested for COVID-19 in the past 30 days
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Only | INFORMED
Number analyzed (Participants) | 121 | 126
Participants
  Tested Tested | 46 | 46
  Not Tested (or missing) | 75 | 80
Statistical Analysis 1: Comparison: Text Messaging Only vs INFORMED; Test type: Superiority; p < 0.05, Mixed Models Analysis; Adjusted for Demographics, COVID-19 Cases Per 100K , Test Access, Social Network, Knowledge, Test Value with random intercepts for participation mode; Odds Ratio (OR) = 0.8378, 95% CI 2-sided [0.4284 to 1.6385] — Adjusted odds ratio

3. Secondary Outcome: COVID-19 Testing Intention
Description: Proportion of participants who "agreed" or "strongly agreed" to the statement "I plan to get tested as often as needed."
Time Frame: Week 16
Population: Participants provided week 16 data
Measure: Count of Participants; unit: Participants
Arm/Group | Text Messaging Only | INFORMED
Number analyzed (Participants) | 116 | 116
Participants
  Agree/Strongly Agree | 84 | 90
  Do not Agree | 32 | 26
Statistical Analysis 1: Comparison: Text Messaging Only vs INFORMED; Test type: Superiority; p < 0.05, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.4306, 95% CI 2-sided [0.6166 to 3.3192] — Adjusted odds ratio

4. Other Pre Specified Outcome: Decisional Conflicts for Getting Vaccinated for COVID-19 Score
Description: Decision conflicts is measured by the 4-item SURE test which asks whether participants: 1) know enough about benefits and harm; 2) clear about which benefits and harms matter most; 3) have enough support/advice to make a choice; and 4) feel sure about the best choice regarding getting vaccinated for COVID-19. Each item is scored either 0 (unsure) or 1 (sure). The total score ranges from 0 to 4. Higher score indicates lower decisional conflicts (or more sure); lower score indicates higher decisional conflicts.
Time Frame: Week 16
Population: Participants who provided the outcome data at follow-up (week 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text Messaging Only | INFORMED
Number analyzed (Participants) | 114 | 114
score on a scale | 3.87 (0.47) | 3.98 (0.13)
Statistical Analysis 1: Comparison: Text Messaging Only vs INFORMED; Test type: Superiority; Mean Difference (Final Values) = 0.08661, 95% CI 2-sided [-0.07311 to 0.2463], Standard Error of Mean 0.08125 — Adjusted for Demographics, COVID Cases Per 100,000 Population, Test Access, Social Network, Knowledge, and Test Value with random intercepts for Dyad and Individual

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Text Messaging Only | INFORMED
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/126
Other Adverse Events (participants affected / at risk) | 0/121 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04893265/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT04893265/ICF_001.pdf